CLINICAL TRIAL: NCT06489249
Title: Role of Inflammation in Vascular Phenotype Associated With E-cigarette Use
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Anna Stanhewicz, PhD, Assistant Professor, University of Iowa
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 202405142
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Electronic Cigarette Use; Endothelial Dysfunction; Inflammation
MeSH Terms: conditions — Vaping; Inflammation | interventions — salicylsalicylic acid; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo then Salsalate (Experimental): Placebo oral table twice daily for 4 days prior to experimental testing followed by 14 day washout period and then salsalate oral tablet 1500mg twice daily for 4 days prior to experimental testing.
  Interventions: Drug: Placebo; Drug: Salsalate 750 MG Oral Tablet [DISALCID]
- Salsalate then Placebo (Experimental): Salsalate oral tablet 1500mg twice daily for 4 days prior to experimental testing followed by 14 day washout period and then placebo oral tablet twice daily for 4 days prior to experimental testing.
  Interventions: Drug: Placebo; Drug: Salsalate 750 MG Oral Tablet [DISALCID]

INTERVENTIONS:
Drug: Placebo — Oral placebo tablet
Drug: Salsalate 750 MG Oral Tablet [DISALCID] — Oral salsalate tablet

SUMMARY:
The use of electronic nicotine delivery systems, or e-cigarettes - colloquially referred to as "vaping" - in the United States has increased exponentially since their introduction to the US market in 2007. Prevalence of ever and current e-cigarette use is highest among teenagers and young adults with 16-28% of this population having reported vaping. While the majority of e-cigarette users are current tobacco smokers, 32.5% of current e-cigarette users are never- or former-smokers, representing a growing population of young adults who exclusively vape. While e-cigarettes have been marketed as a safer alternative to tobacco cigarettes, clinical studies examining these claims are limited. Cardiovascular disease (CVD) is the primary cause of premature death among tobacco cigarette smokers and reductions in vascular endothelial function, a significant predictor of future CVD, are detectible in otherwise healthy young adults who smoke. Despite the explosion in e-cigarette use among young adults, the health effects - especially the effects on mechanisms of vascular function - of these devices remain relatively unexplored. The purpose of this study is to directly asses the mechanistic role of inflammation in this dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 24 years of age
* no history of e-cigarette use (control) OR current with 6 months or more history of e-cigarette use (chronic use).

Exclusion Criteria:

* tobacco cigarette use (current or history of)
* use of stimulant drugs
* skin diseases
* cardiovascular disease
* diagnosed or suspected hepatic or metabolic disease including diabetes
* statin or other cholesterol-lowering medication
* antihypertensive medication
* current pregnancy or breastfeeding
* blood pressure greater than or equal to 140mmHg systolic and/or greater than or equal to 90mmHg diastolic
* allergy to materials used during the experiment
* known allergies to salsalate or other study drugs

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Microvascular endothelial function (Cutaneous conductance, %maximum) following salsalate treatment compared to placebo treatment | a total of 2 times throughout the study (approximately 4 weeks): 1) at the completion of 4 days of oral salsalate treatment, and 2) at the completion of 4 days of placebo treatment
  Endothelium-dependent vasodilation assessed as cutaneous conductance response (cutaneous conductance = local red blood cell flux/mean arterial pressure; %maximum) to local heating of the skin (42 degrees Celcius).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Iowa Bioscience Innovation Facility, Iowa City, Iowa
  - University of Iowa, Iowa City, Iowa

IPD SHARING:
Plan to Share IPD: No